CLINICAL TRIAL: NCT02303665
Title: TCM Multi-channel Interventional Therapy for Assisting Reproduction
Brief Title: Observing the Curative Effect of Assisted Reproduction by TCM Multi-channel Interventional Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Huang Jinzhu, The evaluation of the curative effect onTCM joint treatment intervene in IVF-ET, Chengdu University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012SZ0086
Record Dates: First submitted 2014-11-21; First posted 2014-12-01 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Failure After Assisted Reproductive Technology
Keywords: TCM multi-channel therapy; ART failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- The control group (No Intervention): No Intervention
- The dual therapy group (Experimental): TCM prescriptionⅡof cultivated emotion and assisted reproduction +auricular acupoint therapy.
  Interventions: Other: The dual therapy
- The triple therapy group (Experimental): TCM prescriptionⅡof cultivated emotion and assisted reproduction + auricular acupoint therapy+ retention enema of TCM.
  Interventions: Other: The triple therapy

INTERVENTIONS:
Other: The dual therapy — TCM prescriptionⅡof cultivated emotion and assisted reproduction +auricular acupoint therapy
  Arms: The dual therapy group
Other: The triple therapy — TCM prescriptionⅡof cultivated emotion and assisted reproduction + auricular acupoint therapy+ retention enema of TCM
  Arms: The triple therapy group

SUMMARY:
Objective: To evaluate the curative effect of TCM multi-channel interventional therapy on women with ART Failure; to compare the curative effect of the dual therapy and triple therapy on women with ART Failure; to choose the best TCM interventional therapeutic plan.

Methods: The cases with ART Failure from West China second University Hospital of Sichuan University (West China Women's and Children's Hospital of Sichuan University) meeting the inclusion criteria were randomly divided into three groups: the dual therapy group, the triple therapy group and the control group, compare the natural pregnancy number, the condition during the period of secondary IVF-ET and the improvement of the kidney deficiency, liver depression and blood stasis syndrome among those three groups.

DETAILED DESCRIPTION:
Objective: To evaluate the curative effect of TCM multi-channel interventional therapy on women with ART Failure; to compare the curative effect of the dual therapy and triple therapy on women with ART Failure; to choose the best TCM interventional therapeutic plan.

Methods: The cases with ART Failure from West China second University Hospital of Sichuan University (West China Women's and Children's Hospital of Sichuan University) meeting the inclusion criteria were randomly divided into three groups: the dual therapy group, the triple therapy group and the control group, compare the natural pregnancy number, the condition during the period of secondary IVF-ET and the improvement of the kidney deficiency, liver depression and blood stasis syndrome among those three groups.

The results will show the effect of TCM multi-channel interventional therapy for patients with ART failure

ELIGIBILITY:
Inclusion Criteria:

1. People aged 20 to 45
2. People with IVF - ET indications
3. People from Reproductive Center of West China second University Hospital of Sichuan University (West China Women's and Children's Hospital of Sichuan University) with long plan for IVE - ET Failure and then accept the secondary IVF-ET
4. People who conform to the standard of syndrome differentiation in TCM: kidney deficiency and liver depression and blood stasis
5. People with normal basic sex hormone levels
6. People who have recognized and voluntarily signed the informed consent. NOTICE: People who conform to the above 6 items can be included.

Exclusion Criteria:

1. People don't meet the inclusion criteria
2. The husband with less sperm and weak sperm seriously
3. People who have drug allergy or allergic constitution
4. People with serious primary diseases such as cardiovascular, liver, kidney and hematopoietic system, etc. And mentally disordered patients
5. People who are complicated by acute infectious diseases and organic diseases
6. People have confirmed diagnosis malformed reproductive organs, reproductive system inflammation and tumors upon examination
7. People suffer from hereditary disease which is not suitable for fertility regulated in "maternal and infant health care law"
8. People who have the serious bad habits such as drug use
9. People who have contacted with birth defects rays, poison, drugs to a certain number and being in effect; NOTICE: People who conform to any of the terms above 9 will be ruled out.

Ages: 24 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with sucessful conception | 10 weeks after embryo transplantation

SECONDARY OUTCOMES:
Time to have successful conception | up to 26 weeks
Adverse events | 0, 10, 26 weeks after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Qian Zeng, Study Director — Chengdu University of Traditional Chinese Medicine
Locations (1):
- West China second University Hospital of Sichuan University, Chengdu, Sichuan, China